CLINICAL TRIAL: NCT00446121
Title: The Effect of Inhaled Mannitol on Ciliary Beat Frequency in COPD Patients
Brief Title: Inhaled Mannitol and Ciliary Beat Frequency in COPD Patients
Status: Withdrawn | Type: Observational
Why Stopped: No funding for the project
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 06/Q0410/55
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of the study is to evaluate the effect of mannitol on the cilia's beat frequency (ciliary beat frequency) in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* COPD

Ages: 38 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with COPD
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergei Kharitonov, MD PhD, Principal Investigator — Imperial College London
Locations (1):
- Airway Disease Section, Asthma Lab, Imperial College London, Royal Brompton Hospital, London, United Kingdom